CLINICAL TRIAL: NCT04621383
Title: Effects of Whey Protein Supplementation with Hydrolyzed Collagen Associated with 12 Weeks of Resistance Training on Body Composition, Blood Biomarkers and Muscle Strength in Elderly Women
Brief Title: Effects of Whey Protein Supplementation Collagen Associated to Resistance Training in Older Woman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordination for the Improvement of Higher Education Personnel (Other); Rousselot BVBA (Industry)
Responsible Party: Principal Investigator, Edilson Serpeloni Cyrino, Principal Investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: GPMN2019/02
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia; Collagen Degeneration
Keywords: Resistance training; Sarcopenia; Knee Joint; Cardiometabolic Biomarkers; Lean mass
MeSH Terms: conditions — Sarcopenia | interventions — Whey Proteins; Collagen; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- whey protein plus collagen group (Experimental): Participants received a dose of 30 grams of whey protein plus 20 grams of collagen seven days a week splitted in two servings a day, first one in morning, second one in evening. Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps push-down, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: Whey protein plus collagen
- whey protein plus maltodextrin group (Placebo Comparator): Participants received a dose of 30 grams of whey protein plus 20 grams of maltodextrin seven days a week splitted in two servings a day, first one in morning, second one in evening. Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps push-down, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: Whey protein plus maltodextrin

INTERVENTIONS:
Dietary Supplement: Whey protein plus collagen — This two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 17 weeks. At the beginning of the experiment, two weeks and at the end three weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16), magnetic ressonance imaging (weeks 2 and 17) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.
  Arms: whey protein plus collagen group
Dietary Supplement: Whey protein plus maltodextrin — This two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 17 weeks. At the beginning of the experiment, two weeks and at the end three weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16), magnetic ressonance imaging (weeks 2 and 17) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.
  Arms: whey protein plus maltodextrin group

SUMMARY:
The main purpose of the present study was to investigate the effects of whey protein with collagen hydrolyzed following resistance training on body composition, muscular strength, functional capacity, and plasma-metabolism biomarkers in older women

DETAILED DESCRIPTION:
his two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 17 weeks. At the beginning of the experiment, two weeks and at the end three weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16), magnetic ressonance imaging (weeks 2 and 17) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.

Recruitment was carried out through newspapers, radio advertising, and home delivery of leaflets in the central area and residential neighborhoods. All participants completed health history and physical activity questionnaires and were included in the study if they met the following inclusion criteria: 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction that would prevent them from performing the prescribed exercise or exercise testing associated with the study, not receiving hormonal replacement therapy, and completed a previous 8-week RT programParticipants underwent a diagnostic graded exercise stress test with a 12-lead electrocardiogram reviewed by a cardiologist and were released with no restrictions for participation in this investigation.

A blinded researcher was responsible for generating random numbers for participant allocation. Both groups were submitted to the same RT program and all participants completed the experiment. Written informed consent was obtained from all participants after a detailed description of investigation procedures was provided. This investigation was conducted according to the Declaration of Helsinki and was approved by the local University Ethics Committee The Shapiro Wilk test will be used to test data distribution. Data will be presented as means, standard deviation, and z-score. The student's independent t-test and chi-square test were will be used to compare groups regarding the general characteristics and clinical/medical history (categorical variables). Two-way analysis of variance (ANOVA) for repeated measures will be used to assess between group comparisons. The effect size (ES) will be calculated to verify the magnitude of the differences by Cohen's d, where an ES of 0.20-0.49 will be considered as small, 0.50-0.79 as moderate, and ≥ 0.80 as large(41). The Z-score of the percentage changes (from pre- to post-training) of the raw data for each parameter will be calculated, as well as a total Z-score, derived from all the components. To verify the differences between groups in total Z-scores, an independent T test will be also applied. For all statistical analyses, significance was accepted at P < 0.05. The data will be analyzed using SPSS software version 20.0 (SPSS, Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

60 years old or more, physically independent, free from cardiac or orthopedic dysfunction that would prevent them from performing the prescribed exercise or exercise testing associated with the study, not receiving hormonal replacement therapy, and completed a previous 8-week RT program. In this study, only women with SO were included. SO was defined as a body fat mass ≥ 35% combined with appendicular lean soft tissue (ALST) less than <15.02 kg, assessed by dual x-ray energy absorptiometry (DXA). Participants underwent a diagnostic graded exercise stress test with a 12-lead electrocardiogram reviewed by a cardiologist and were released with no restrictions for participation in this investigation.

Exclusion Criteria:

All subjects not participating in 85% of the total sessions of training or withdraw

-

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Change in body composition | baseline and after 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) (Lunar Prodigy) was used to assess lean mass and fat mass and its segments. The total skeletal muscle mass (SMM) was estimated by the predictive equation proposed by Kim et al. (Kim et al., 2004). The results are presented in kg.
Change in Muscular strength | baseline and after 12 weeks
  Maximal dynamic strength was evaluated using the 1RM test assessed on chest press, knee extension, and preacher curl exercises performed in this exact order. Testing for each exercise was preceded by a warm-up set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warm-up was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load in three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the last resistance lifted in which the subject was able to complete only one single maximal execution
Change in knee cartilage | baseline and after 12 weeks
  Magnetic resonance imaging was used to access the thickness of knee cartilage in multiaxial protocol. the total cartilage was measured by a trained tecnician on images. The results are presented in mm.

SECONDARY OUTCOMES:
Change in Total cholesterol | Measurements of serum levels of total cholesterol were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
  Measurements of serum levels of total cholesterol were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in high-density lipoprotein (HDL-C) | baseline and after 12 weeks
  Measurements of serum levels of high-density lipoprotein were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in triglycerides | baseline and after 12 weeks
  Measurements of serum levels of triglycerides were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in low-density lipoprotein | baseline and after 12 weeks
  For the determination of LDL-c was used the Friedewald equation: LDL-c=TC - (HDL-c + TG / 5).
Change in glucose | baseline and after 12 weeks
  Measurements of serum levels of glucose (GLU) were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring).
Change in insulin | baseline and after 12 weeks
  Insulin was determined by the chemiluminescence method (LIASON equipment)
Change in HOMA-IR | baseline and after 12 weeks
  The Homeostasis Assessment Model (HOMA-IR) was calculated by the formula: Insulin fasting (μUI / mL) x Glucose fasting (mmol / L) / 22.5.
Change in blood pressure | baseline and after 12 weeks
  Resting BP assessment was performed using automatic, oscillometric equipment (Omron - 7113). Participants attended the laboratory on three different days and, during each visit, remained seated at rest for 10 min with the cuff of the equipment in place on the right arm. Subsequently, several BP measurements were performed at one-minute intervals in order to obtain three consecutive measurements where the difference in systolic BP (SBP) and diastolic BP (DBP) readings differed by no more than 4 mmHg. The average of the three measurements for each day was averaged across the three visits.
Change in body mass | baseline and after 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale, with subjects wearing light workout clothing and no shoes.
Change in height | baseline and after 12 weeks
  Height was measured using a stadiometer to the nearest 0.1 cm while subjects were standing without shoes.
Change in body mass index | baseline and after 12 weeks
  Body mass index was calculated as the body mass in kilograms divided by the square of the height in meters.
Change in waist circumference | baseline and after 12 weeks
  We also collected data on waist circumference (WC), using a flexible and inelastic tape measure. WC was obtained at the midpoint between the last rib and the iliac crest at the time of expiration. Two measurements were used to measure each circumference. In situations in which the difference between the measurements was greater than 0.5 cm a third measurement was performed, with the value of the median being adopted as reference. All measurements were performed by the same evaluator.
Change in hip circumference | baseline and after 12 weeks
  We also collected data on hip circumference, using a flexible and inelastic tape measure. HC was measured in the region of greater perimeter between the waist and the thigh. Two measurements were used to measure each circumference. In situations in which the difference between the measurements was greater than 0.5 cm a third measurement was performed, with the value of the median being adopted as reference. All measurements were performed by the same evaluator.
Dietary intake | baseline and after 12 weeks
  Food consumption were assessed by the 24-hour dietary recall method applied on two non-consecutive days of the week, with the aid of a photographic record taken during an interview. The homemade measurements of the nutritional values of food and supplementation were converted into grams and milliliters by the online software Virtual Nutri Plus for diet analysis. Some foods were not found in the program database and therefore items were added from food tables.
Change in inflammatory markers | baseline and after 12 weeks
  Tumor Necrosis Factor -α (TNF-α) and Interleukin-6 (IL-6) were determined by enzyme-linked immunosorbent assay (ELISA), according to the specifications of the manufacturer and performed in a microplate reader Perkin Elmer, model EnSpire (USA). All samples were determined in duplicate to guarantee the precision of the results. The results are presented in picograms per milliliter (pg/ml).
Change in hepatic markers | baseline and after 12 weeks
  Aspartate aminotrasferase(AST), Alanine aminotransferase(ALT) , were determined by enzimatic method (IFCC Technology: Cobas 6000 - Roche) and and Gamma glutamyl transferase(γ-GT) were determined by colorimetric enzimatic method(IFCC Technology: Cobas 6000 - Roche) according to the specifications of the manufacturer, All samples were determined in duplicate to guarantee the precision of the results. The results are presented in units by liter (U/L).
Change in C-reactive protein (CRP) | baseline and after 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligrams per decilitre (mg/dL).
Change in Uric acid | baseline and after 12 weeks
  Uric acid , were determined by colorimetric enzimatic method (Technology: Cobas 6000 - Roche) according to the specifications of the manufacturer, All samples were determined in duplicate to guarantee the precision of the results. The results are presented in miligrams by deciliter (mg/dL).
Change in Urea | baseline and after 12 weeks
  Uric acid, were determined by kinetic method (Technology: Cobas 6000 - Roche) according to the specifications of the manufacturer, All samples were determined in duplicate to guarantee the precision of the results. The results are presented in miligrams by deciliter (mg/dL).
Change in Creatinine | baseline and after 12 weeks
  Creatinine, were determined by kinetic colorimetric method (Technology: Cobas 6000 - Roche) according to the specifications of the manufacturer, All samples were determined in duplicate to guarantee the precision of the results. The results are presented in miligrams by deciliter (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Edilson S Cyrino, PhD., Study Director — Universidade Estadual de Londrina
Locations (1):
- Rodrigo dos Reis Fernandes, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Sardinha LB, Lohman TG, Teixeira PJ, Guedes DP, Going SB. Comparison of air displacement plethysmography with dual-energy X-ray absorptiometry and 3 field methods for estimating body composition in middle-aged men. Am J Clin Nutr. 1998 Oct;68(4):786-93. doi: 10.1093/ajcn/68.4.786. PMID 9771855
- [Background] Kim J, Heshka S, Gallagher D, Kotler DP, Mayer L, Albu J, Shen W, Freda PU, Heymsfield SB. Intermuscular adipose tissue-free skeletal muscle mass: estimation by dual-energy X-ray absorptiometry in adults. J Appl Physiol (1985). 2004 Aug;97(2):655-60. doi: 10.1152/japplphysiol.00260.2004. Epub 2004 Apr 16. PMID 15090482